Potential for Cortisol Suppression With the Use of High Volume Nasal Mometasone Irrigations in Varying Dosages.

NCT03979209

8/10/2021

Statistical Analysis Plan

An a priori analysis using G\*3.0.10 Power was performed in order to determine adequate sample size. Using a Cohen's D of 1.0, alpha of 0.05 and power of 0.95, sample size was determined to be 13. Pre- and post-treatment morning cortisol serum levels were compared using a match paired, dependent sample Student's t-test. Significance was established at P < 0.05. All data acquired during this study were de-identified to protect patient privacy, and identifying information was only available to the principal investigator.